CLINICAL TRIAL: NCT04400084
Title: Ex Vivo Study of Drugs Transfer Across the Placenta
Brief Title: Using Cotyledon Perfusion to Study Drugs Transfer Across the Placenta
Acronym: DRUGS-PTP
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190817
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Normal Pregnancy
Keywords: Placenta; Drug; Transplacental transfer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant mothers: Pregnant mothers who have a normal pregnancy
  Interventions: Other: Placenta perfusion

INTERVENTIONS:
Other: Placenta perfusion — Placenta perfusion in double closed circuit, during 3 hours

SUMMARY:
Drug prescriptions are usual during pregnancy however women and their fetuses still remain an orphan population with regard to drugs efficacy and safety clinical studies. Most xenobiotics diffuse through the placenta and some of them can alter fetus development resulting in structural abnormalities, growth or functional deficiencies. The aim of the study is to study the drug transfer using human placenta after delivery.

DETAILED DESCRIPTION:
For ethical reasons, pregnant woman are not included in clinical trials so that data regarding safety and efficacy of many drugs are scarce. It is known that xenobiotics across the placental barrier but studies regarding quantity and mechanisms of this transfer remain insuffisant. Among the different methodologies to evaluate drug transfer, perfusion of human cotyledon is one of the most relevant ones. The two sides of the cotyledon, fetal and maternal ones, are perfused within the hour after delivery with EARLE medium in a double closed circuit. The studied drug (it can be any drug given to pregnant mothers) and antipyrine (the control molecule) are added at the beginning of the three hours perfusion realized at 37°C, with maternal flow rate of 12ml/min and fetal one of 6ml/min. Samples are collected along the perfusion and the drugs dosage will be done in the pharmacology department of Cochin Hospital. Tissues of the cotyledon will be also collected to study the proteins, and ARNs expressed. The drug concentrations will be analyzed by calculating fetal to maternal concentrations ratios and a fetal transfer rate (fetal drug quantity on total drug quantity at the end of the perfusion). Then modelling on Monolix software will be done to estimate the transfer constants across the two compartments. Modelling will allow to estimate the interindividual variability and to test covariables like sex, gestation duration, genetics, or protein expression. Proteins will be studied by an appropriated method (western blot, or proteomic analysis). The genetics study will consist in candidate gene approach. Polymorphisms will be chosen in genes coding for transporters or enzymes or their regulators.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women older than 18 years,
* patient with social security or health insurance,
* from the 24th week of amenorrhea,
* patient who has given her consent,

Exclusion Criteria:

* Maternal pathologies pre-existing pregnancy :

  * diabetes-like vascular disease,
  * arterial hypertension,
  * known prothrombotic pathology, history of venous thrombosis or pulmonary embolism,
  * maternal serology HIV+, BHV+, CHV+ and syphilis,
* Pregnancy and fetal pathologies :

  * pre-eclampsia,
  * delayed growth in utero (can affect placental circulation),
  * gestational diabetes without insulin,
  * fetal malformation,
  * known genetic pathology,
* Patient under tutorship or curatorship, or not speaking french,
* Patient who has not given her consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women who give birth in the Port-Royal maternity (Paris)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Fetal transfer rate | At 180 minutes (end of the perfusion)
  Quantity of drug transferred into fetal compartment/ quantity of drug in the two compartments *100

SECONDARY OUTCOMES:
Ratio of concentrations | At 180 minutes (end of the perfusion)
  Fetal concentration / maternal concentration *100

CONTACTS AND LOCATIONS:
Locations (1):
- CIC Port-Royal-Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schneider H, Panigel M, Dancis J. Transfer across the perfused human placenta of antipyrine, sodium and leucine. Am J Obstet Gynecol. 1972 Nov 15;114(6):822-8. doi: 10.1016/0002-9378(72)90909-x. No abstract available. PMID 4676572
- [Background] Hutson JR, Garcia-Bournissen F, Davis A, Koren G. The human placental perfusion model: a systematic review and development of a model to predict in vivo transfer of therapeutic drugs. Clin Pharmacol Ther. 2011 Jul;90(1):67-76. doi: 10.1038/clpt.2011.66. Epub 2011 May 11. PMID 21562489
- [Background] Preta LH, Bouazza N, Foissac F, Froelicher L, Urien S, Dauvilliers A, Dinnall A, Buth V, Benaboud S, Treluyer JM, Lui G. Comparison of human transplacental transfer of escitalopram, sertraline and paroxetine: an ex vivo cotyledon perfusion study. Placenta. 2025 Aug;168:150-158. doi: 10.1016/j.placenta.2025.06.015. Epub 2025 Jun 24. PMID 40580785